CLINICAL TRIAL: NCT04538781
Title: AMBULATE VASCADE MVP Same Day Discharge Retrospective Registry
Status: Completed | Type: Observational
Sponsor: Cardiva Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL 0617
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Same Day Discharge: Patients undergoing a-fib ablation procedures who were closed with VASCADE MVP and were discharged the same day.
  Interventions: Device: VASCADE MVP VVCS

INTERVENTIONS:
Device: VASCADE MVP VVCS — The VASCADE MVP Venous Vascular Closure System (VVCS) is indicated for the percutaneous closure of femoral venous access sites while reducing time to ambulation, total post-procedure time, time to hemostasis, and time to discharge eligibility in patients who have undergone catheter-based procedures utilizing 6 - 12F inner diameter (maximum 15F OD) procedural sheaths, with single or multiple access sites in one or both limbs.

SUMMARY:
A multi-center, retrospective, single arm post market registry to evaluate procedural outcomes data using the Cardiva VASCADE MVP Venous Vascular Closure System (VVCS) for the management of the femoral venotomy after catheter-based atrial fibrillation interventions with or without another arrythmia performed via 6-12F procedural sheaths with single or multiple access sites per limb for patients who are discharged the same day.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. Underwent catheter-based ablation for atrial fibrillation with or without another arrythmia.
3. VASCADE MVP was the only closure device utilized.
4. Were discharged the same calendar day as the index procedure.
5. Completed a SOC follow-up > 7 days post-procedure.

Exclusion Criteria:

1. Any additional procedure(s) involving femoral arterial or venous access in either limb within the SOC follow up period as defined by each site (minimum 7 days post-procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects 1) treated for A-Fib with or without another arrythmia via catheter ablation 2) who received VASCADE MVP with no other vascular closure device and 3) were discharged the same calendar day during the retrospective date range.
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Freedom from next day access site closure-related complications requiring hospital intervention | 1 day
  Primary Performance Outcome
rate of major venous access site closure-related complications | ≥7 days
  Major Complication rate

SECONDARY OUTCOMES:
Freedom from next day procedure-related complications requiring hospital intervention | 1 day
  Secondary Performance Outcome
Freedom from access site closure-related complications requiring hospital intervention through standard of care follow up contact | ≥7 days
  Secondary Performance Outcome
minor venous access site closure-related complications | ≥7 days
  Minor Complication rate

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Coastal Cardiology, San Luis Obispo, California
  - MedStar Washington, Washington D.C., District of Columbia
  - Lahey Clinic, Burlington, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No